CLINICAL TRIAL: NCT02713542
Title: Autologous Conditioned Plasma (ACP) Intra-articular (IA) Injections for Knee Osteoarthritis (OA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 004
Record Dates: First submitted 2016-02-04; First posted 2016-03-18 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- Autologous Conditioned Plasma (ACP) (Experimental): 3 Intra-articular (IA) injections at 1 week intervals
  Interventions: Device: ACP
- Normal Saline (NS) (Placebo Comparator): 3 NS Intra-articular (IA) injections at 1 week intervals
  Interventions: Other: Placebo

INTERVENTIONS:
Device: ACP — Autologous Conditioned Plasma
  Arms: Autologous Conditioned Plasma (ACP)
Other: Placebo — Three Normal Saline IA injections of 3-8 mL at 1-week intervals.
  Other Names: Normal Saline
  Arms: Normal Saline (NS)

SUMMARY:
This study is primarily investigating the effectiveness of Autologous Conditioned Plasma (ACP) Intra-articular (IA) in patients with Osteoarthritis (OA) in the knee.

DETAILED DESCRIPTION:
This study is a prospective, multi center randomized double blind, two arm study.

90 subjects will be randomized to receive injections of either Autologous Conditioned Plasma Intra-articular or the control.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 18 to 70 years of age.
2. The subject presents with complaints of continued pain of primary knee for at least 6 weeks.
3. The subject has documented radiographs evidence of Osteoarthritis (OA) in the tibio-femoral or patella-femoral compartment of the target knee (Kellgren-Lawrence Grades II-III), using radiographs performed within 24 weeks of screening.
4. The subject has a WOMAC pain score of at least 8 out of 20 and at least moderate pain (a score of 2) for at least 2 questions on activities

Exclusion Criteria:

1. Grade I and IV on the knee Kellgren-Lawrence grading scale
2. Subject has clinically 3+ effusion of the target knee (stroke test grading system).
3. Subject has significant (> 10⁰) valgus or varus deformities as evidenced by standard of care X-ray.
4. Subject has had systemic or IA injection of corticosteroids in any joint within three months prior to screening.
5. Viscosupplementation in any joint in the past six months.
6. Subject has an increased risk for post- procedure bleeding (e.g., bleeding disorder or taking anticoagulants except low-dose aspirin).
7. Subject had prior open surgery on the target knee within 12 months or knee arthroscopy within 6 months
8. Subject has inflammatory disease of either knee other than OA.
9. Subject with underlying medical conditions that could interfere with the evaluation of the outcome.
10. Subject with positive pregnancy test, or breast feeding.
11. Subject with plans to participate in other clinical trial involving medical or surgical intervention in the next 12 months.
12. Subject with any condition (including cognitive impairment) that, in the opinion of the investigator, might interfere with the evaluation of the study objectives.
13. Subject has rheumatoid arthritis or gout
14. Subject has a history of or a current infection at the affected joint.
15. Subject with plans to undergo any elective orthopedic surgery in the next 12 months.
16. Subject requires pain management therapy (with the exception of acetaminophen) not related to the target knee.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-07; Primary Completion 2018-07-02 (Actual); Study Completion 2018-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Smith, MD, Principal Investigator — Columbias Orthopedic Group
Locations (4):
- United States (4):
  - Rush University Medical Center, Chicago, Illinois
  - MedSport University of Michigan Sports Medicine, Ann Arbor, Michigan
  - Columbia Orthopedic Group, Columbia, Missouri
  - Hawkins Foundation, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 126 patients were evaluated and 90 were treated at four sites
Pre-assignment Details: A total of 36 patients were excluded before randomization to groups due to not meeting Inclusion/Exclusion criteria.
Period: Overall Study
Arm/Group | Autologous Conditioned Plasma (ACP) | Normal Saline (NS)
Started | 60 | 30
Completed | 42 | 24
Not Completed | 18 | 6
Not completed — Use of prohibited medication | 14 | 5
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Autologous Conditioned Plasma (ACP): Three Intra-articular injections of ACP in knee at 1 week intervals
- Control: Normal Saline (NS): Three Intra-articular injections of NS in knee knee at 1 week intervals
- Total: Total of all reporting groups
Arm/Group | Experimental: Autologous Conditioned Plasma (ACP) | Control: Normal Saline (NS) | Total
Number analyzed (Participants) | 60 | 30 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (10.3) | 50.6 (10.9) | 51.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 15 | 49
  Male | 26 | 15 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 15 | 46
  Not Hispanic or Latino | 23 | 13 | 36
  Unknown or Not Reported | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 32 | 16 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 23 | 14 | 37
Region of Enrollment [Number; unit: participants]
  United States | 60 | 30 | 90
WOMAC pain score of at least 8 [Count of Participants; unit: Participants] | 60 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores Measured by Western Ontario and McMaster Universities Index (WOMAC) Survey
Description: The WOMAC Pain score will be used to measure outcome, the score ranges from 0 to 20. The higher the score indicates greater pain.
Time Frame: 6 month visit
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Autologous Conditioned Plasma: 3 Intra-articular injections of ACP in knee at 1 week intervals
- Normal Saline: 3 Intra-articular injections of NS in knee at 1 week intervals
Arm/Group | Autologous Conditioned Plasma | Normal Saline
Number analyzed (Participants) | 42 | 24
units on a scale | 3.98 [0 to 17] | 5.54 [0 to 18]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Autologous Conditioned Plasma (ACP) | Normal Saline (NS)
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/30
Other Adverse Events (participants affected / at risk) | 32/60 | 21/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Conditioned Plasma (ACP) (N=60) | Normal Saline (NS) (N=30)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
eye disorder (Eye disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Virus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flu (General disorders) | 2 (2) | 0 (0)
Pain in Target knee (Musculoskeletal and connective tissue disorders) | 11 (17) | 8 (8)
Pain (not in target knee) (Musculoskeletal and connective tissue disorders) | 13 (16) | 10 (10)
Joint effusion (Musculoskeletal and connective tissue disorders) | 7 (9) | 1 (1) — swelling in knee
Stiffness in target knee (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Tendinitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Atrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint noises in target knee (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Decreased range of motion in target knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Parasthesia (Nervous system disorders) | 1 (1) | 0 (0) — not device procedure or disease related
Paralysis (Nervous system disorders) | 1 (1) | 0 (0) — not device , procedure or disease related
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary pain (Renal and urinary disorders) | 1 (1) | 0 (0)
cold (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Injection site pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) — not related to device, procedure or disease
Skin CA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hematoma in target knee (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the Clinical Trial Agreement between sponsor and PI it states, "Institution and clinical Investigator may not publish or publicly present the results of the study without the prior written approval of sponsor."

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT02713542/Prot_SAP_000.pdf